CLINICAL TRIAL: NCT05239559
Title: Feasibility and Acceptability Followed by Effectiveness of Bubble Continuous Positive Airway Pressure for Treatment of Bangladeshi Children With Severe Pneumonia
Brief Title: Feasibility and Acceptability Followed by Effectiveness of bCPAP for Treatment of Bangladeshi Children With Severe Pneumonia
Acronym: Child-bCPAP
Status: Completed | Type: Observational
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Edinburgh (Other); NIHR Global Health Research Unit on Respiratory Health (RESPIRE) (Unknown); Director General of Health Services, Bangladesh (Unknown)
Responsible Party: Sponsor
Other Study IDs: PR-18049
Record Dates: First submitted 2018-10-16; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-12

CONDITIONS: Feasibility
Keywords: Childhood; Severe Pneumonia; Hypoxaemia; bubble continuous positive airway pressure; Feasibility and acceptability
MeSH Terms: conditions — Pneumonia; Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- bubble CPAP arm: Oxygen will be delivered by Bubble CPAP device, which will have three components:
  1. Continuous gas flow into the circuit: The gas flow rate required to generate CPAP is usually 5-10 L/min.
  2. A nasal interface connecting the child's airway with the circuit: short nasal prongs are generally used to deliver nasal CPAP. They must be carefully fitted to minimize leakage of air (otherwise, CPAP will not be achieved) .
  3. An expiratory arm with the distal end submerged in water to generate end-expiratory pressure: in bubble CPAP, the positive pressure is maintained by placing the far end of the expiratory tubing in water. The pressure is adjusted by altering the depth of the tube under the surface of the water.
  Interventions: Device: Bubble CPAP oxygen delivery device

INTERVENTIONS:
Device: Bubble CPAP oxygen delivery device — In Bubble CPAP, pressurized oxygen from an oxygen cylinder is delivered to the nasopharynx of the baby. An underwater tube (expiratory arm) that acts as a blow off valve is interposed between the oxygen source and the baby. Adjusting the height of the water column above the exit of the tube can regulate the pressure in the system and the amount of CPAP delivered to the baby. The constant bubbling of gas through the blow off mechanism delivers the bubbling CPAP effect. Oxygen may be delivered by nasal prongs inserted into the nostril of child.
  The system has three components:
  1. Continuous gas flow into the circuit: The gas flow rate required to generate CPAP is usually 5-10 L/min.
  2. A nasal interface connecting the child's airway with the circuit:
  3. An expiratory arm with the distal end submerged in water to generate end-expiratory pressure.
  The source of oxygen will be either an oxygen concentrator or cylinder, central distribution through pipelines.

SUMMARY:
Background: Feasibility and acceptability of bubble continuous positive airway pressure (CPAP) were not evaluated in childhood severe pneumonia in developing countries at a larger scale.

Objective:

1. To describe prevailing structural and functional conditions and other operational challenges in nontertiary hospitals in Bangladesh that would need to be addressed in order to introduce bubble CPAP as part of the management of children with severe pneumonia enabling a successful interventional trial.
2. To develop and test bubble CPAP training materials of relevance to clinical staff providing care for children with severe pneumonia in district general hospitals.
3. To determine the prevalence of hypoxaemia among hospitalised children with severe pneumonia in non-tertiary/district hospitals, current practices with regard to management and clinical outcome, to support power calculations of a future interventional trial of bubble CPAP for children with severe pneumonia.
4. To document the early experience, particularly the feasibility and acceptability of introducing bubble CPAP in selected non-tertiary/district hospitals.

Methodology:

Feasibility/demonstration phase will be done as an internal pilot in 2 hospitals. Current treatment practice, facilities, and operational challenges will be evaluated for the introduction, clinical use and maintenance of bubble CPAP.

Outcome:

1. To describe the structural and functional conditions and operational challenges that may influence the introduction of bubble CPAP.
2. To have bubble CPAP training materials that can be delivered cheaply and repeatedly to a level of comprehension of staff providing care to children with pneumonia in district general hospitals in Bangladesh.
3. A quantitative analysis of the incidence of hypoxaemia among hospitalised children with severe pneumonia, current management practices and clinical outcomes.
4. A qualitative assessment of the feasibility of introducing bubble CPAP.

Number of children to be enrolled: 20 children in 2 hospitals as an internal pilot (i.e. 10 in each hospital)

Main inclusion criteria: Age between 2 months and 24 months with severe pneumonia and hypoxemia and guardian/parent gives written informed consent to participate in the study.

Statistical Analysis: For feasibility and acceptability study, a descriptive analysis will be performed.

Study duration: 44 months

ELIGIBILITY:
INCLUSION CRITERIA

* Staff:

  * Staff (medical and nursing) employed at the two selected hospitals with duties that include care of children with pneumonia
  * Staff who agree to participate and give written informed consent
* Children for assessment of hypoxaemia in pneumonia and outcomes:

  * Age between 2 - 24 months
  * Attend one of the two study hospitals for the assessment of pneumonia by hospital clinician.
  * Pneumonia defined by WHO criteria
* Children receiving bubble CPAP:

  * Age between 2 - 24 months.
  * Diagnosis of pneumonia by a hospital clinician together with hypoxaemia (SpO2<90%).
  * Parent/guardian gives informed consent to participate in the study

EXCLUSION CRITERIA

* Hospital staff:

  o There will be no exclusion criteria
* Children for assessment of hypoxaemia in pneumonia and outcomes, and children receiving bubble CPAP:

  * Known congenital heart disease, asthma, pulmonary TB and other chronic respiratory disorders

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 2-24 months having hypoxaemia in pneumonia (Pneumonia defined by WHO criteria)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The structural, functional and operational challenges will be described | 44 month
  Human resources, Supply chain, logistics equipment maintenance, power failure, disconnection of oxygen with local complications will be identified.
To have bubble CPAP training materials that can be delivered cheaply and repeatedly to a level of comprehension of staff providing care to children with pneumonia in district general hospitals in Bangladesh | 44 month
  The training module, Standard Operating Procedure, treatment algorithm will be provided to the hospital staff. Hands-on training will be done.
A quantitative analysis of the incidence of hypoxaemia among hospitalised children with severe pneumonia, current management practices and clinical outcomes | 44 month
  Prevalence, management, mortality, referral, discharge, hospital stay, oxygen therapy duration of severe pneumonia cases will be identified.
Feasibility and acceptability of introducing bubble CPAP | 44 month
  Challenges related to the introduction of bCPAP, enrollment, patient management with follow-up recording, human resources, respiratory support will be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Md. Mohammod J Chisti, PhD, Principal Investigator — Senior Scientist
Locations (2):
- Bangladesh (2):
  - Institute of Child and Mother Health, Dhaka
  - 250 bedded General hospital, Kustia

IPD SHARING:
Plan to Share IPD: No
After the end of the study, data will be analyzed as ter the defined data analysis plan on the protocol. Study results will be shared with other researchers by journal publications, conferences proceedings and dissemination programs